Appendix – II: Informed Consent Form

Research topic: Association of salivary amino acid with oral squamous cell carcinoma

identified by liquid chromatography mass spectrometry.

Principle Investigator: Dr. DipayanMojumder

The aim of this consent form is to inform you all the necessary information, which will help you

to take decision whether you will participate in this research or not.

**Aim and Procedure:** 

The aim of the study is to find out the association of salivary amino acid levels with oral

squamous cell carcinoma (OSCC). The study will be conducted at Oral and Maxillofacial Surgery

Department of Bangabandhu Sheikh Mujib Medical University Patient with histologically

confirmed OSCC will be enrolled as cases in the study by purposive convenient sampling

technique to achieve the desired number. Approximately same number of the healthy individuals

will be taken as control group for comparison. Then the saliva will be taken from the OSCC

patient and from the control group. After taking in the sterile container and ensuring proper

environment saliva sample will be carried to Designated Reference Institute for Chemical

Measurements (DRICM), Science lab, Dhanmondi for analysis by liquid chromatography-mass

spectrometry (LC-MS) machine. By this machine, the levels of 6 specific amino acids (Alanine,

Valine, Glycine, Phenylalanine, Isoleucine, Lysine) will be measured. The data obtained from

each individual will be recorded in predesigned data collection sheet separately. If you are

agreeing to participate in this research program, the responsible doctor will inform you in detail.

#### Risk of this Research:

Risk of this research is minimum. But, this risk will be addressed by proper treatment. If any problem arises related to the biopsy procedure or due to any step of this research activity, you will get the whole treatment in free of cost.

#### Advantage of participation in this research program:

You might be benefited by participating in this research program. The problems related to OSCC will be addressed by medication, operative procedure and follow up visit.

### **Alternative way:**

You will get the appropriate treatment in this hospital even after not participating in research program.

#### **Cost:**

You will not have to pay or you will not be paid for participating in this research program.

#### **Confidentiality:**

During and after research program confidentiality would be maintained strictly. An ID number will be given to you and that will be helpful to the research program. All thepapers belong to this ID number will be locked in office. Personal matter will not be used for analysis, producing article and release. Only the involved investigator will know all these and nobody will get their information.

# **Voluntary participation:**

Your participation in this research program is absolutely voluntary. You can either deny participation or leave the research program at any time. That will not affect your treatment process. Your legal right will not be harmed by signing this form.

### **Queries:**

Please ask if you have any question. We will try our best to answer. If any question arises in your mind in the future, please contact with the researcher **Dr. DipayanMojumder**, Oral and Maxillofacial Surgery Department, Block- A, BSMMU.

# **Agreement:**

I am satisfied by the counseling of the responsible doctor for this research program who will do my physical examination. I could understand that participation in this research program is voluntary and I could leave this research program at any time without anyobligation. I have gone through all the above condition/ was read in front of me and Iam agreeing to participate in this research program voluntarily.

| <u>Informed by:</u> | <u>Participant:</u> | Witness: |
|---------------------|---------------------|----------|
| Name: | Name: | Name: |
| Sign: | Sign: | Sign: |
| Date: | | |